CLINICAL TRIAL: NCT02254317
Title: Dose-dependent Effect of Grape Seed Extract (GSE) on Glucose Control in People With Impaired Glucose Tolerance
Brief Title: Dose-dependent Effect of Grape Seed Extract on Glucose Control in People With Impaired Glucose Tolerance
Acronym: GSE3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2014-074
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Impaired Glucose Tolerance
Keywords: Impaired Glucose Tolerance; Oral Glucose Tolerance Test; Grape Seed Extract
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0 mg placebo (Placebo Comparator): Not containing GSE (Placebo)
  Interventions: Dietary Supplement: 0 mg placebo
- 300 mg GSE (Active Comparator): Containing 300 mg of GSE
  Interventions: Dietary Supplement: 300 mg GSE
- 600 mg GSE (Active Comparator): Containing 600 mg of GSE
  Interventions: Dietary Supplement: 600 mg GSE
- 900 mg GSE (Active Comparator): Containing 900 mg of GSE
  Interventions: Dietary Supplement: 900 mg GSE

INTERVENTIONS:
Dietary Supplement: 0 mg placebo — Not containing GSE (Placebo)
  Other Names: Placebo Comparator
  Arms: 0 mg placebo
Dietary Supplement: 300 mg GSE — 300 mg GSE
  Other Names: Active Comparator1
  Arms: 300 mg GSE
Dietary Supplement: 600 mg GSE — Containing 600 mg of GSE
  Other Names: Active Comparator2
  Arms: 600 mg GSE
Dietary Supplement: 900 mg GSE — Containing 900 mg of GSE
  Other Names: Active Comparator3
  Arms: 900 mg GSE

SUMMARY:
The objective is to identify the lowest effective dose of Grape Seed Extract (GSE) on glucose control in people with impaired glucose tolerance (IGT).

DETAILED DESCRIPTION:
The proposed study is a single-center, placebo-controlled, randomized, 4-arm, crossover study that identify the lowest effective dose of GSE on glucose control in people with impaired glucose tolerance.

A planned sample size of 20 will be recruited into the study. This study will require one initial screening visit, pre-study visit, and 4 Oral Glucose Tolerance Test Days (OGTT) Days. This study will take 4-6weeks per subject to complete.

The trial will initiate with one screening visit, which will last for about 3-4 hours where the subjects' height, weight, BMI, waist circumference, fasting blood glucose, blood pressure and heart rate will be measured and a survey related to general eating, health and exercise habits will be completed. OGTT procedure will be performed to confirm IGT.

If willing and eligible to participate, a 3-day food record (2 weekdays and 1 weekend) will be given at the screening visit and collected on the following pre-study Visit to assess subject's baseline dietary intake and pattern. Also, subjects will be instructed to follow a relatively low polyphenolic-diet at least 7 days prior to the first OGTT Day and for the duration of the study. A dinner meal will be provided the day before the OGTT Day to control the second meal effect from food and beverage intake of the night before the OGTT Day.

Subjects will arrive at the center in a fasting state for at least 10 hours, well hydrated and rested. Each OGTT Day will require blood draws throughout the visit. After evaluation of subject's health status (via anthropometric, vital sign and blood glucose measurements and in-person interview), a registered nurse will place a catheter in subject's arm for the purpose of multiple blood sample collections and take the initial blood draw (baseline: -1h) in the fasting state. 3 test capsules with 0 mg GSE, 300 mg GSE, 600 mg GSE or 900 mg GSE (in forms of: 3 placebo, 2 placebo & 1 GSE, 1 placebo & 2 GSE or 3 GSE. Each GSE capsule containing 300 mg GSE) will be served. Thereafter, timers will be started and a glucose test drink (75g glucose mixed with 250ml water) will be given right after the 0h blood sampling (1 h after the consumption of capsules). Subject will be instructed to finish the drink in 5 minutes (min). From this point forward, blood sample will be collected at 30 min, 1h, 2hand 3h for assessment of changes in metabolic markers. The sequence of receiving the capsules treatment at each visit will be randomly assigned based on computer generated sequences.

OGTT Day visits will be placed at least 3 days apart as well.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 to 65 years old male/female
* Body Mass Index (BMI) less than 35kg/m2
* Fasting blood sugar between 100-125 mg/dL
* Confirmed impaired glucose tolerance (IGT) upon 2 hr OGTT screening test (≥ 140 mg/dL < 200mg/dL)
* Non-smoker
* No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Not taking any medications or dietary supplements that would interfere with outcomes of the study.

Exclusion Criteria:

* Past smokers: abstinence for less than 2 years
* Men and women who smoke
* Men and women with known or suspected food intolerance, allergies or hypersensitivity to the study materials or closely related compound or any their stated ingredients.
* Men and women known to have/diagnosed with diabetes mellitus
* Men and women who have fasting blood glucose concentrations ≥126 mg/dL
* Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries.
* Men and women with cancer other than non-melanoma skin cancer in previous 5 years.
* Men and women who are taking medication or dietary supplements that may interfere with the outcomes of the study; e.g., antioxidant supplements, anti-inflammation, lipid lowering medication. Subjects may choose to go off dietary supplements (requires 30 days washout).
* Men and women who have donated blood within 3 months of the screening visit and blood donors/participants for whom participation in this study will result in having donated more than 1500 milliliters of blood in the previous 12 months.
* Substance (alcohol or drug) abuse within the last 2 years.
* Excessive coffee and tea consumers (> 4 cups/day)
* Unstable weight: gained or lost weight +/- 5 lbs in previous 3 months
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study and women who are lactating.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2015-06-27 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in plasma metabolic markers over 4 hour Oral Glucose Tolerance Test (OGTT) after administration of GSE capsules (containing 300mg, 600mg or 900mg Grape seed extract) compared to 0 mg placebo. | 4 hr
  plasma metabolic markers over 4 hour Oral Glucose Tolerance Test (OGTT)

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Eunyoung Park, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No